CLINICAL TRIAL: NCT03946904
Title: Clinical Study of Laser Analgesia in Cavity Preparations
Brief Title: Clinical Study of Laser Analgesia in Cavity Preparations Using the Er,Cr:YSGG Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Laser Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-CHEN-101
Record Dates: First submitted 2019-05-03; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Tooth Pain
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- preconditioning (Experimental): Patients with towo similar size lesions of either Class I or class v cavities selected as subjects. in the same appointment, both cavities are prepared by the Er'Cr:YSGG. The lesion in this case was prepared with low power setting to start and is aimed at applying low level laser therapy (LLLT) first before using high power.
  Interventions: Device: Er,Cr:YSGG Laser
- no preconditioning (Experimental): Patients with towo similar size lesions of either Class I or class v cavities selected as subjects. in the same appointment, both cavities are prepared by the Er'Cr:YSGG.the lesion in this case was prepared with high power laser setting first to ablate the enamel, dentin, and caries.
  Interventions: Device: Er,Cr:YSGG Laser

INTERVENTIONS:
Device: Er,Cr:YSGG Laser — Patients with towo similar size lesions of either Class I or class v cavities selected as subjects. in the same appointment, both cavities are prepared by the Er'Cr:YSGG. one lesion was prepared with high power laser setting first to ablate the enamel, dentin, and caries. the other lesion was prepared with low power setting to start and is aimed at applying low level laser therapy (LLLT) first before using high power.
  Other Names: Iplus laser

SUMMARY:
Not much has been done in research to explain the clinical benefit of laser cavity preparation without the use of injection anesthetic. The Author of this study sought to show the science behind the "no shot, no pain" in restorative dentistry using an Er,Cr:YSGG laser Patients with two similar size lesions of class I or class V cavities selected as subjects. In the same appointment, both cavities are prepared by the Er,Cr:YSGG. One lesion was prepared with one high power laser setting to ablate the enamel, dentin, and caries. The other lesion was prepared with a low power setting to start and is aimed at applying low level laser therapy (LLLT) before using the high power setting to ablate enamel, dentin, and caries. A visual analog scale (VAS) was used for the patient to analyze how comfortable each laser technique was. An Analysis of Variance (ANOVA) was used.

DETAILED DESCRIPTION:
The principal objective of this study is to prove the phenomenon of laser analgesia. Traditionally before a cavity preparation is performed, the doctor will use local anesthetic (Needle Injection) before using rotary instrument to do a cavity preparation. The study involves using the Er,Cr=YSGG Laser to perform cavity preparation without giving any injection anesthesia. VAS (Visual Analog Scale) will be used to have patients rate the laser cavity preparation procedure to show there is laser analgesia. On each patient subject that has two similar size cavities of the same classification, either Class I or Class V, on similar teeth. Two different laser protocols will be used. One includes Low Level Laser Therapy (LLLT) to condition the pulp producing analgesia before using higher power to perform the cavity prep. The other protocol will skip the LLLT setting and prepare the cavity with the higher power to perform the cavity prep. The design of the study is to find out if there is laser analgesia and if LLLT makes a difference in providing better analgesia. The VAS forms from each procedure will be used to show there is laser analgesia and potentially cavity preparations can be performed by using the laser without the need to give injection anesthesia first. 48 patients will be included in this study.

Treatment. Preconditioning and cavity preparation are done using the Er:Cr:YSGG laser, Waterlase MD (mfg: Biolase Technology Inc, Irvine CA), and the gold hand piece with an MG6 fiber tip, trunk fiber, contra-angle hand piece. Preconditioning. Preconditioning is preformed using laser desensitization. One tooth will be randomly selected, and preconditioning will be performed using LLLT on the tooth with minimal tooth ablation. The LLLT settings that will be used for preconditioning are 0.25 Watts, 50 Hz, 0% water, 0% air, H mode. Following this a fiber-optic tip will be aimed perpendicular to the surface of the cervical portion of the tooth, ensuring that a 2mm distance will be maintained between the end of the fiber optic tip and the surface. The fiber-tip will be used to generate a 2mm line. The cavity on the second tooth will be prepared for without laser preconditioning. Lesion Preparation - small preparations. Small preparations are to be performed as follows. The Waterlase MD is set to 4.5W, 15 Hz, 65% air, and 60% water and the cavity is prepared according to the preferred technique. If patients indicate sensitivity, the procedure will be halted, patients fill out the VAS form and anesthetic will be offered. For patients who refuse anesthetic, the procedure will be continued at the same settings. Lesion Preparation - small to medium preparations. Small to medium preparations will be performed as follows. The Waterlase MD will be set to 2W, 15 Hz, 65% air, and 60% water and the cavity will be prepared according to the preferred technique. If patients indicate sensitivity, the procedure will be halted, patients fill out the VAS form and anesthetic will be offered. For patients who refuse anesthetic, the procedure will be continued at the same settings.

Restoration. Overall VAS Score. Up to 3 intra-operative VAS measurements are recorded. If a patient feels even the slightest amount of pain during the procedure, they will be instructed to raise their hand and the treatment will be paused. The patient is then asked to fill in the VAS form before the procedure will be continued. After conclusion of the cavity preparation, patients will be asked to mark one last VAS rating indicating the overall pain of the procedure. Patients that do not raise their hand throughout the entirety of the procedure will be given an overall VAS rating of zero. Data for each patient will be recorded and analyzed in this way.

The VAS scale will be presented to the patients using a standard explanation (zero, indicating no pain at all, to 100, representing the 'worst pain patient had ever felt'). Patients will be asked to place a vertical line on the VAS scale to indicate his/her discomfort status. They are encouraged to stop the treatment if they encounter any pain. The number of hand raises, as defined by the protocol, will be recorded and analyzed (small and medium/large preparations are analyzed separately), represent the number of times during the procedure the patient felt sufficient discomfort to stop the procedure. VAS data will be assessed by the following assumptions: The 'lower' the average score, the 'better' the mode of treatment. Once the patient marks their vertical line on the scale, a precise measurement, in millimeters, was taken from the "zero" line of the VAS scale to where the patient marked their line.

ELIGIBILITY:
Inclusion Criteria:

* You are an adult 19-65 years of age who had at least two cavity preparations of the same type, with the same approximate size lesion.
* No language barriers
* Not Pregnant
* Immune system is not compromised (No bronchitis, no sinus infection, no ear infection, or any other infection of any type ect…)
* No Heart Disease
* No high blood pressure
* No teeth amalgam restorations were in close proximity to the lesion.
* Requiring at least two cavity preparations of the same type, with the same approximate size of lesion (minimum 1mm diameter x 1mm depth).

Exclusion Criteria:

* Children
* Pregnant women
* Immune compromised patients
* Patients with heart disease
* High blood pressure
* Cardiac arrhythmia
* Patients whose teeth amalgam restorations were in close proximity to the lesion
* Decay that has reached the pulp where potential for root canal therapy
* Patients of different language difficulty

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Clinical Study of Laser Analgesia in Cavity Preparations using the Er,Cr:YSGG Laser | 1 year
  Preconditioning the cavity with LLLT will result in effective analgesia and the cavity preparation will be virtually painless. Overall VAS Score: Up to 3 intra-operative VAS measurements will be recorded. If a patient felt any pain at all during the procedure, they were instructed to raise their hand and the treatment would be paused. The patient was then asked to fill in the VAS form and then the procedure continued. After the conclusion of the cavity preparation, the patients were asked to fill in one last VAS form rating the overall pain of the procedure. Patients that did not raise their hand throughout the entirety of the procedure were given an overall VAS rating of zero. Data for each patient will be recorded and analysed in this way.

CONTACTS AND LOCATIONS:
Overall Officials: William H Chen, doctor, Principal Investigator — Chen Laser Institute
Locations (1):
- Chen Laser Institute, Granite City, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03946904/Prot_000.pdf